CLINICAL TRIAL: NCT03032445
Title: Potential Impacts of Beer on Post-Race Ultramarathon Athletes
Brief Title: Beer for Endurance Exercise Recovery
Acronym: BEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Jeremy Joslin, MD, Associate Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beer Trial
Record Dates: First submitted 2017-01-12; First posted 2017-01-26 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hyponatremia
Keywords: Body Water/physiology; Hyponatremia/etiology; Physical Exertion/physiology; Running/physiology; Sodium/blood; Ethanol
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcoholic beer (Experimental): At least 6% alcohol content
  Interventions: Other: Alcoholic Beer
- Non alcoholic beer (Placebo Comparator): Less than 0.5% alcohol content
  Interventions: Other: Non alcoholic beer

INTERVENTIONS:
Other: Alcoholic Beer — Subject will be asked to consume alcoholic beer within 30 minutes. Subject will be monitored for 60 minutes at commencement of study beverage.
  Arms: Alcoholic beer
Other: Non alcoholic beer — Subject will be asked to consume non alcoholic beer within 30 minutes. Subject will be monitored for 60 minutes at commencement of study beverage.
  Arms: Non alcoholic beer

SUMMARY:
Athletes who are participating in the Keys100 Ultramarathon event in Key West, FL are eligible, based on inclusion criteria, to participate in this research study that is seeking to determine whether supplementation of beer (alcohol) immediately following a long distance ultramarathon race can positively impact exercise-associated hyponatremia [EAH].

ELIGIBILITY:
Inclusion Criteria:

* Completed informed consent
* Ability to read and speak English language
* Age 21 years or older
* Not considered a vulnerable population, such as pregnant (by history) or cognitively impaired.
* Able to tolerate needle exposure for blood draw
* Willing to drink alcoholic or nonalcoholic beer
* Willing not to eat or drink other than the study fluid during 1 hour study period
* Participating in 100 mile or 50 mile race
* To participate in the controlled part of the study the individual must have fully completed either the 100 mile or the 50 mile race.

Exclusion Criteria:

* Under age 21 years
* Vulnerable population, such as pregnant (by history) or cognitively impaired
* Subjects who are alcohol-naive (i.e first exposure to alcohol)
* Subjects with known familial and/or genetic backgrounds at higher risk for the development of alcohol dependence
* Subjects should not be seeking treatment for alcohol or drug abuse
* Subjects who are in general high risk for abuse such as those completing or participating in alcohol or drug abuse programs
* Subjects who have had a sustained period of abstinence, with history of heavy drinking problems, while living in the community

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-21 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
Changes in sodium level pre and post intervention | One hour

SECONDARY OUTCOMES:
Measurement of urine output | One hour
Number of participants with abnormal laboratory values | One hour
Level of cognition | Within one month of intervention
  Cognitive level determined by assessment of clock drawing test.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Joslin, MD, Principal Investigator — SUNY Upstate Medicial University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No